CLINICAL TRIAL: NCT06318065
Title: Prognostic Factors Impacting Surgical Resection Outcomes in Patients With Brain
Brief Title: Surgical Resection Outcomes in Patients With Brain Metastasis
Status: Recruiting | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B-ER111-370
Record Dates: First submitted 2024-02-25; First posted 2024-03-19 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-02

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
While many studies have investigated the prognostic factors for patients undergoing surgical resection for primary brain tumors, decision-making for patients with brain metastasis (BM) is more complex because of their higher burden of comorbidities compared to those with primary brain tumors. In addition, although various prognostic indicators have been identified to predict prognosis in several types of cancer, such as the neutrophil-to-lymphocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR), prognostic nutritional index (PNI), and systemic immune-inflammation index (SII), limited studies have yet determined which group of patients would yield beater survival outcome after surgical resection for BM. This study aimed to investigate the impact of patient and perioperative characteristics and prognostic indicators on survival outcome of patients undergoing surgical resection of BM.

ELIGIBILITY:
Inclusion Criteria:

1. patients with Clinical diagnosis of brain metastasis
2. patients who underwent craniotomy surgery for brain metastasis

Exclusion Criteria:

1. patients with insufficient data for associated factors
2. patients who underwent stereotactic biopsy for brain metastasis
3. patients who did not undergo craniotomy surgery for brain metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients newly diagnosed with BM due to various primary cancers who underwent surgery at our institution
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
survival outcome of patients undergoing surgery for brain metastasis | From date of surgery until the date of death from any cause, whichever came first, assessed up to 100 months
  overall survival of patients
Functional outcome of patients undergoing surgery for brain metastasis | from date of surgery until 6 months after surgery ordate of death from any cause, whichever came first
  change of preoperative and postoperative modified rankin scale

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Shun Lee, M.D., Study Chair — National Cheng Kung Univsersity Hospital
Locations (1):
- Jung-Shun Lee, Tainan, None Selected, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided